CLINICAL TRIAL: NCT00004062
Title: Restoration of Radioiodine Uptake in Thyroid Carcinoma: A Clinical Trial
Brief Title: Azacitidine to Restore Thyroid Function in Patients With Persistent or Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lucille P. Markey Cancer Center at University of Kentucky (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067262; UKMC-9700053; NCI-T99-0045
Record Dates: First submitted 1999-12-10; First posted 2004-06-04 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2004-05

CONDITIONS: Head and Neck Cancer
Keywords: stage IV papillary thyroid cancer; stage IV follicular thyroid cancer; recurrent thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid Neoplasms | interventions — Azacitidine; Triiodothyronine; Iodine-131

INTERVENTIONS:
Drug: azacitidine
Drug: liothyronine sodium
Radiation: iodine I 131

SUMMARY:
RATIONALE: Azacitidine may help thyroid cancer cells regain the ability to take up iodine. This would allow the cancer to be detected and treated by radioactive iodine.

PURPOSE: Phase I trial to study the effectiveness of azacitidine to restore thyroid function in treating patients who have persistent or metastatic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the ability of azacitidine to restore iodine uptake by dedifferentiated thyroid cancer, enabling detection and treatment with iodine I 131 in patients with metastatic follicular or papillary thyroid cancer. II. Evaluate different doses and schedules of azacitidine administration to determine an optimally effective combination for restoration of iodine I 131 uptake with acceptable toxicity in this patient population. III. Determine the efficacy of azacitidine plus iodine I 131 in this patient population.

OUTLINE: This is a dose escalation study of azacitidine. Patients undergo a control phase consisting of oral liothyronine sodium twice daily on weeks 1-4 and a low iodine diet on weeks 4-7. At week 6, patients receive a scan dose of iodine I 131 followed by whole body scanning over 5 days. Beginning at week 7, patients undergo a treatment phase consisting of oral liothyronine sodium twice daily for 3 weeks, azacitidine subcutaneously daily for 10 or 20 days (weeks 7-11) and a low iodine diet on weeks 8-11. During week 11, patients undergo additional whole body scanning over 5 days followed by a therapeutic dose of iodine I 131. Patients achieving successful therapy receive 5 additional doses of azacitidine. Cohorts of 4 patients receive escalating doses of azacitidine until demonstrable radioiodine uptake is seen or the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 8 patients experience dose limiting toxicity. Patients are followed weekly for 8 weeks.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Radiologically confirmed persistent or metastatic follicular or papillary thyroid cancer following total thyroidectomy and radioiodine ablation therapy Metastatic disease confirmed histologically or cytologically or by elevated thyroglobulin levels No radioiodine uptake by whole body scanning Stable iodine contamination from radiologic contrast material within the past 10 months allowed, if absence of current contamination demonstrated by less than 80 micrograms of iodine in a 24 hour urine collection

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT/SGPT no greater than 2.5 times upper limit of normal (ULN) Bilirubin no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN OR Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: At least 4 weeks since prior levothyroxine Any prior therapy for restoration of radioiodine uptake allowed, if unsuccessful and did not exceed treatment schedules planned for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ain, MD, Study Chair — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky, United States